CLINICAL TRIAL: NCT01350622
Title: Efficacy of PENNSAID® for Pain Management in the Emergency Department
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never initiated
Sponsor: University of Utah (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 49065
Record Dates: First submitted 2011-04-29; First posted 2011-05-10 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Pain; Ankle Sprain
Keywords: pain management
MeSH Terms: conditions — Pain; Ankle Injuries; Agnosia | interventions — Diclofenac; diclofenac hydroxyethylpyrrolidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pennsaid (Experimental): Active Pennsaid and oral placebo
  Interventions: Drug: PENNSAID
- Oral Diclofenac (Active Comparator): Oral diclofenac and placebo lotion (2.3% DMSO solution)
  Interventions: Drug: Diclofenac hydroxyethylpyrrolidine

INTERVENTIONS:
Drug: PENNSAID — active treatment with PENNSAID and oral placebo. Subjects will apply 40 drops of Pennsaid to the affected ankle joint once, and will take a single placebo pill.
  Arms: Pennsaid
Drug: Diclofenac hydroxyethylpyrrolidine — active treatment oral Diclofenac and PENNSAID placebo. Patients will take a single 50mg dose of oral diclofenac and will apply 40 drops of placebo lotion (2.3% DMSO) to the affected ankle once.
  Arms: Oral Diclofenac

SUMMARY:
The primary objective of this study is to compare the pain relieving effect and speed of onset of PENNSAID to that of standard oral diclofenac under double blind conditions using a growth curve approach to pain measurement. The investigators will test the hypothesis that PENNSAID will provide more rapid pain relief than oral diclofenac during the ED visit. The secondary goal of the proposed work is to discover and model the onset and course of pain relief during the emergency department (ED) visit.

ELIGIBILITY:
Inclusion:

-We will include ED patients presenting with an acutely painful ankle sprain for which NSAIDs constitute standard of care pain management.

The following will be excluded:

* Those with lacerations, bites, burns
* any head trauma
* pregnant
* anyone with a pre-existing chronic pain condition
* inflammatory intestinal disorders such as Crohn's disease or ulcerative colitis
* anyone regularly using another NSAID or anti-coagulation medication
* anyone who has experienced asthma after NSAID use
* compromised cognitive abilities
* a significant co-morbidity that will compromise participation
* had joint replacements
* known hypersensitivity to diclofenac or allergic responses to NSAIDs as a class
* active stomach and/or duodenal ulceration or gastrointestinal bleeding
* anyone admitted with severe active bleeding
* recent heart surgery
* severe liver or renal insufficiency
* prisoner
* mentally disabled patients
* wards of the state
* cognitive or decisional impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Change in pain score | Measure at 5 minute intervals for the duration of the ER visit
  Compare the pain relieving effect and speed of onset of PENNSAID to that of standard oral diclofenac.

SECONDARY OUTCOMES:
pain trajectory model | nine months
  The secondary goal of the proposed work is to discover and model the onset and course of pain relief during the ED visit

CONTACTS AND LOCATIONS:
Overall Officials: Richard Chapman, PhD, Study Director — University of Utah; Virgil Davis, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Baer PA, Thomas LM, Shainhouse Z. Treatment of osteoarthritis of the knee with a topical diclofenac solution: a randomised controlled, 6-week trial [ISRCTN53366886]. BMC Musculoskelet Disord. 2005 Aug 8;6:44. doi: 10.1186/1471-2474-6-44. PMID 16086839
- [Background] Chapman CR, Donaldson GW, Davis JJ, Bradshaw DH. Improving individual measurement of postoperative pain: the pain trajectory. J Pain. 2011 Feb;12(2):257-62. doi: 10.1016/j.jpain.2010.08.005. Epub 2011 Jan 15. PMID 21237721
- [Background] Moen MD. Topical diclofenac solution. Drugs. 2009;69(18):2621-32. doi: 10.2165/11202850-000000000-00000. PMID 19943711
- [Background] Pritchard PH, Brindley DN. Studies on the ethanol-induced changes in glycerolipid synthesis in rats and their partial reversal by N-(2-benzoyloxyethyl)norfenfluramine (benfluorex). J Pharm Pharmacol. 1977 Jun;29(6):343-9. doi: 10.1111/j.2042-7158.1977.tb11332.x. No abstract available. PMID 18570
- [Background] Galer BS. A comparative subjective assessment study of PENNSAID(R) and Voltaren Gel(R), two topical formulations of diclofenac sodium. Pain Pract. 2011 May-Jun;11(3):252-60. doi: 10.1111/j.1533-2500.2010.00420.x. Epub 2010 Sep 20. PMID 20854305
- [Background] Roth SH, Shainhouse JZ. Efficacy and safety of a topical diclofenac solution (pennsaid) in the treatment of primary osteoarthritis of the knee: a randomized, double-blind, vehicle-controlled clinical trial. Arch Intern Med. 2004 Oct 11;164(18):2017-23. doi: 10.1001/archinte.164.18.2017. PMID 15477437
- [Background] Rupp T, Delaney KA. Inadequate analgesia in emergency medicine. Ann Emerg Med. 2004 Apr;43(4):494-503. doi: 10.1016/j.annemergmed.2003.11.019. PMID 15039693
- [Background] Todd KH, Ducharme J, Choiniere M, Crandall CS, Fosnocht DE, Homel P, Tanabe P; PEMI Study Group. Pain in the emergency department: results of the pain and emergency medicine initiative (PEMI) multicenter study. J Pain. 2007 Jun;8(6):460-6. doi: 10.1016/j.jpain.2006.12.005. Epub 2007 Feb 15. PMID 17306626
- [Background] Towheed TE. Pennsaid therapy for osteoarthritis of the knee: a systematic review and metaanalysis of randomized controlled trials. J Rheumatol. 2006 Mar;33(3):567-73. PMID 16511925
- [Background] Tugwell PS, Wells GA, Shainhouse JZ. Equivalence study of a topical diclofenac solution (pennsaid) compared with oral diclofenac in symptomatic treatment of osteoarthritis of the knee: a randomized controlled trial. J Rheumatol. 2004 Oct;31(10):2002-12. PMID 15468367
- [Background] Hui X, Hewitt PG, Poblete N, Maibach HI, Shainhouse JZ, Wester RC. In vivo bioavailability and metabolism of topical diclofenac lotion in human volunteers. Pharm Res. 1998 Oct;15(10):1589-95. doi: 10.1023/a:1011911302005. PMID 9794502